CLINICAL TRIAL: NCT03398369
Title: Advanced Imaging and Inflammatory Markers to Define Mechanisms of Response to CRT
Brief Title: Mechanistic Clinical Trial of Advanced Imaging for CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kenneth Bilchick, MD, Associate Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UVAMRICRTTRIAL
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): CMR-Guided CRT
  Interventions: Diagnostic Test: CMR/CTA Guidance for CRT
- Control (No Intervention): Standard CRT

INTERVENTIONS:
Diagnostic Test: CMR/CTA Guidance for CRT — The intervention is the use of CMR and CTA to determine the optimal pacing site in the left ventricle for cardiac resynchronization therapy (CRT) and guide left ventricular lead placement.
  Arms: Intervention

SUMMARY:
This is a mechanistic clinical trial with randomization to guidance for the CRT procedure using cardiac magnetic resonance (CMR) and computed tomography angiography (CTA) versus a standard procedure.

DETAILED DESCRIPTION:
At baseline, patients will have CMR, CTA, echocardiography, blood testing, and cardiopulmonary exercise testing. They will also complete a heart failure questionnaire. In patients randomized to CMR guidance for the CRT procedure, LV lead placement will be guided by the MRI information related to scar, activation and anatomy. Patients will have follow-up assessments at 6 and 12 months. There will also be clinical follow-up for survival free of appropriate ICD therapies over 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic systolic HF
2. LVEF 35% or less
3. Guideline-based class I or II indication for CRT

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnancy
3. Presence of metal embedded in the body due to prior accident or injury, as documented by skull films or other imaging
4. Cerebral aneurysm clips
5. Cochlear implants
6. Other metallic implants known to be contraindications to CMR (does not include pacemakers and ICDs)
7. Severe claustrophobia
8. Acute kidney injury
9. Acute renal failure or chronic kidney disease with GFR < 45 cc/min/1.73m2
10. Liver transplant
11. Gadolinium allergy
12. >10% premature ventricular contraction (PVC) burden; and 13) estimated >10% atrial fibrillation (AF) burden based on available clinical data.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Left ventricular end-systolic volume (LVESV) improvement | One Year
  Change in LVESV with cardiac resynchronization therapy (CRT)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Bilchick, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No